CLINICAL TRIAL: NCT01415323
Title: Agitation in the Acute Psychiatric Department
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Bergen (Other); University of Oslo (Other); Deakin University (Other)
Responsible Party: Sponsor
Other Study IDs: Acute agitation
Record Dates: First submitted 2011-07-06; First posted 2011-08-11 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Mental Disorders
Keywords: Emergency services, psychiatric; Psychomotor agitation; Suicide; Violence
MeSH Terms: conditions — Mental Disorders; Psychomotor Agitation; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected for storage and analyses both at admittance and discharge from the psychiatric acute department.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acutely admitted psychiatric in-patients

SUMMARY:
Agitation is associated with a number of acute psychiatric conditions, and frequent in acute psychiatric admissions. It is associated with violence towards others, and strongly associated with in-patient suicides.

The main aims of the study are to assess different clinical presentations of agitation at admittance, and to assess the consequences of these different clinical presentations during the first three days of the stay.

DETAILED DESCRIPTION:
The patients are assessed with three rating scales (Components of agitation, The PANSS-EC, The Brøset Violence Checklist) measuring agitation at admittance and day three thus providing a measurement of the differences during three days of in-patient stay. Therapeutic measures and interventions taken are assessed daily with a 18-item checklist. Threatening and violent incidents are recorded with The SOAS-R.

Blood samples for immunological parameters are taken at admittance and discharge giving opportunity to assess changes through the acute psychiatric condition. Urine and blood samples are taken at admittance to assess substance use and medications.

The patients are assess with two self-rating VAS-scales at discharge assessing the suicidal intentions they have had during the stay, aspects of clinical history and assessment for personality disorders.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive acutely admitted in-patients are asked for participation.

Exclusion Criteria:

* Patients not willing to sign informed consent form.
* Patients not speaking English or Norwegian.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acutely admitted psychiatric in-patients from a defined catchment area.
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
the number of violent or threatening incidents the first three days of inpatient stay measured with The Staff Observation Aggression Scale - Revised (SOAS-R) with positive scorings of incidents with a severity score >8. | Up to 4 years.

SECONDARY OUTCOMES:
the degree of suicidal intention the first three days of inpatient stay measured with the 10 item self-rating VAS-scale administered at discharge from the acute department. | Up 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Arne E Vaaler, PhD, MD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- St Olavs University Hospital, Department of Acute Psychiatry Østmarka, Trondheim, Norway

REFERENCES:
- [Result] Sallaup TV, Vaaler AE, Iversen VC, Guzey IC. Challenges in detecting and diagnosing substance use in women in the acute psychiatric department: a naturalistic cohort study. BMC Psychiatry. 2016 Nov 17;16(1):406. doi: 10.1186/s12888-016-1124-y. PMID 27855664
- [Result] Nakken EI, Grinde F, Vaaler A, Drange OK, Brodtkorb E, Saether SG. Epilepsy and other seizure disorders in acute psychiatric inpatients. BMC Psychiatry. 2021 Dec 15;21(1):626. doi: 10.1186/s12888-021-03619-y. PMID 34911471
- [Derived] Krane-Gartiser K, Vaaler AE, Fasmer OB, Sorensen K, Morken G, Scott J. Variability of activity patterns across mood disorders and time of day. BMC Psychiatry. 2017 Dec 19;17(1):404. doi: 10.1186/s12888-017-1574-x. PMID 29258468